CLINICAL TRIAL: NCT02755506
Title: Study on The Value of Endobronchial Ultrasound Elastography in The Diagnosis of Thoracic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Liang_An, Director of respiratory medicine, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S2016-020-01
Record Dates: First submitted 2016-04-15; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Thoracic Lesions
Keywords: Ultrasound elastography; Thoracic lesions; EBUS-TBNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with thoracic lesions (Experimental): Patients with thoracic lesions is going to undergo endobronchial ultrasound elastography followed by endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA).
  Interventions: Device: endobronchial ultrasound elastography

INTERVENTIONS:
Device: endobronchial ultrasound elastography — Before endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), patients will undergo the examination of endobronchial ultrasound elastography

SUMMARY:
The study aims to evaluate the role of endobronchial ultrasound elastography in differentiated diagnosis of benign and malignant thoracic lesions

DETAILED DESCRIPTION:
Ultrasound elastography has been gradually used in clinic with the rapid development of ultrasonic technique,and presents a promising application prospect in differentiated diagnosis of benign and malignant disease.The aim of the study is to evaluate the accuracy of endobronchial ultrasound elastography in the diagnosis of thoracic lesions.

Conventional ultrasound and ultrasound elastography are respectively used to examine thoracic lesions before aspiration,then the images are saved as video clips. Features of conventional ultrasound and parameters of ultrasound elastography are analysed and recorded by skilled worker. The investigators define the pathological results of EBUS-TBNA combined with results of six months follow-up as the "Gold Standard". The receiver operator characteristic curves are drawn to obtain area under the Curve (AUC) and the best diagnostic threshold values of each parameters. According to the best cutoff values, the investigators respectively calculate the accuracy, sensitivity, specificity, odds product of each parameters, and then compare them with each other to evaluate the value of ultrasound elastography

ELIGIBILITY:
Inclusion Criteria:

* Hilar/mediastinal lymph lesions with a short axis more than 1 cm on thoracic computed tomography( CT) scan and/or positron emission tomography-computed tomography (PET-CT)
* With normal Coagulation function
* With normal cardio pulmonary function and be able to tolerate bronchoscopy
* No syphilis,acquired immune deficiency syndrome(AIDS) and other infectious diseases
* Willing and able to give written informed consent

Exclusion Criteria:

* Unable to lie in bed
* Allergy to narcotics such as lidocaine.
* Suffering from cardiovascular and cerebrovascular disease, severe lung liver and kidney dysfunction, or after drug treatment cannot maintain the normal.
* With abnormal Coagulation function or take anticoagulant drugs within the previous week.
* Hematological abnormalities, fever or highly suspected active tuberculosis patients.
* Women in the menstrual period.
* Excessive anxiety and can not tolerate bronchoscopy.
* Other conditions that are not suitable for inclusion in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Elastography strain ratio | six months
  Elastography strain ratios were calculated between selected area of the lesions and the surrounding normal tissues.Then ROC curve was drawn to obtain the best diagnostic threshold value.According to the best cutoff value, the diagnostic accuracy,sensitivity and specificity of strain ratio were calculated.The pathological results of EBUS-TBNA combined with results of long-term follow-up were defined as the gold standard.
Elasticity score | six months
  Elasticity scores were obtained by analyzing elastography images.Scores:1-2: benign;3-4: malignant lesions. The sensitivity and specificity of elastography for the diagnosis of malignant thoracic lesions were calculated on the basis of above-specified criteria. The pathological results of EBUS-TBNA combined with results of long-term follow-up were defined as the gold standard.
Elastography area ratio | six months
  Elastography area ratios were defined as following:areas as blue pixels/lesion areas as region of interest pixels.Then ROC curve was drawn to obtain the best diagnostic threshold value.According to the best cutoff value, the diagnostic accuracy,sensitivity and specificity of area ratio were calculated.The pathological results of EBUS-TBNA combined with results of long-term follow-up were defined as the gold standard.

SECONDARY OUTCOMES:
Comparison of value of endobronchial ultrasound elastography in differentiated diagnosis of thoracic lesions with that of conventional ultrasound. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Liang-an Chen, MD,PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Because of personal privacy, the research-related individual participant data do not intend for public sharing.